CLINICAL TRIAL: NCT03266159
Title: A Phase I/II Open-Label, Dose Escalation Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics, and Clinical Activity of GSK525762 Plus Trametinib in Subjects With Small Cell Lung Cancer and Ras-Mutated Solid Tumors
Brief Title: A Dose Escalation Study to Investigate the Safety, Pharmacokinetics (PK), Pharmacodynamics (PD), and Clinical Activity of GSK525762 Plus Trametinib in Subjects With Solid Tumors
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study withdrawn before active to fully evaluate impact of changing practice in target population.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 204673
Record Dates: First submitted 2017-08-25; First posted 2017-08-30 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Solid Tumours
Keywords: Dose escalation; Small cell lung cancer; Trametinib; GSK525762; Ras-mutations; BET inhibitor
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — trametinib

STUDY DESIGN:
Intervention Model Description: A sequential combined therapy of GSK525762 plus trametinib will be given to the subjects. Subjects will receive escalating doses in part 1 and the dose combination selected at the end of part 1 will be provided in part 2.
Masking Description: This will be an open-label study. Hence, masking will not be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1: Subjects receiving GSK525762 + trametinib (Experimental): Eligible subjects will receive doses of GSK525762 with a starting dose of 40 milligrams (mg), or 60 mg in combination with trametinib with a starting dose of 1 mg or 1.5 mg or 2 mg, administered orally once daily. Dose escalation will continue until the maximally-tolerated dose combination (MTC) is reached. Once the MTC is reached, subjects will be enrolled in expansion cohort and will receive a fixed dose combination.
  Interventions: Drug: GSK525762 Besylate tablets; Drug: Trametinib tablets
- Part 2: Subjects with SCLC receiving GSK525762+ trametinib (Experimental): Eligible subjects with small cell lung cancer (SCLC) will receive their Part 2 dose as the dose combination of GSK525762 with trametinib selected at the end of Part 1.
  Interventions: Drug: GSK525762 Besylate tablets; Drug: Trametinib tablets
- Part 2: Subjects with RMCRC receiving GSK525762+ trametini (Experimental): Eligible subjects with Ras-mutated colorectal cancer (RMCRC) will receive their Part 2 dose as the dose combination of GSK525762 with trametinib selected at the end of Part 1.
  Interventions: Drug: GSK525762 Besylate tablets; Drug: Trametinib tablets
- Part 2: Subjects with RMNSCLC receiving GSK525762+ trametinib (Experimental): Eligible subjects with Ras-mutated non small cell lung cancer (RMNSCLC) will receive their Part 2 dose as the dose combination of GSK525762 with trametinib selected at the end of Part 1.
  Interventions: Drug: GSK525762 Besylate tablets; Drug: Trametinib tablets
- Part 2: Subjects with RMPAC receiving GSK525762+ trametinib (Experimental): Eligible subjects with Ras-mutated pancreatic adenocarcinoma (RMPAC) will receive their Part 2 dose as the dose combination of GSK525762 with trametinib selected at the end of Part 1.
  Interventions: Drug: GSK525762 Besylate tablets; Drug: Trametinib tablets
- Part 2: Subjects with RAST receiving GSK525762+ trametinib (Experimental): Eligible subjects with Ras-pathway activated solid tumors (RAST) will receive their Part 2 dose as the dose combination of GSK525762 with trametinib selected at the end of Part 1.
  Interventions: Drug: GSK525762 Besylate tablets; Drug: Trametinib tablets

INTERVENTIONS:
Drug: GSK525762 Besylate tablets — GSK525762 Besylate film coated tablets will be available as a 20 mg tablet strength, yellowish pink in color, round and biconvex with no markings. It will be administered with 240mL of liquid.
Drug: Trametinib tablets — Trametinib film coated tablets will be available as 0.5 mg and 2 mg dose strengths. Trametinib 0.5 mg will be yellow colored, modified oval, biconvex, tablets with 'GS' debossed on one face and 'TFC' on the opposing face.
  Trametinib 2 mg will be pink colored, round, biconvex tablets with 'GS' debossed on one face and 'HMJ' on the opposing face. Doses will be taken at least 1 hour before or at least 2 hours after a meal.

SUMMARY:
GSK525762 is a novel inhibitor of bromodomain and extraterminal (BET) proteins. Trametinib is a potent inhibitor of the mitogen-activated protein kinase proteins (MEK1 and MEK2). GSK525762 and trametinib are critical for growth and survival of tumor cells. This will be the first study demonstrating the synergistic effect of BET inhibitor and MEK inhibitor administered together against tumor cell growth. This study aims to evaluate the safety, tolerability, PK, PD, and preliminary efficacy of combination of GSK525762 and trametinib when administered concomitantly to subjects with small cell lung cancer (SCLC) and rat sarcoma virus oncogene homolog (Ras) mutated solid tumors. The study will be conducted in two parts; part 1 will consists of dose escalation and dose expansion cohorts and part 2 will consists of four disease specific cohorts (SCLC, Ras-mutated adenocarcinoma [RMAC] of the colon [Ras-mutated colorectal cancer {RMCRC}] and/or rectum, Ras-mutated non small cell lung cancer [RMNSCLC], Ras-mutated pancreatic adenocarcinoma [RMPAC]) and an optional "basket" cohort (Ras-pathway activated solid tumors [RAST]). Part 1 will focus on selection of the Part 2 dose based on safety/tolerability, PK, PD, and efficacy. Part 2 will investigate the overall response rate and clinical response. The total duration of study will be approximately three years (nine to twelve months for part 1 and two years for part 2). Approximately 138-156 subjects will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent provided.
* Males and females 18 years old and greater, at the time of signing the informed consent.
* Histologically- or cytologically confirmed diagnosis of one of the following; Part 1 dose escalation cohorts: Advanced (metastatic or non-resectable) SCLC with any mutational status, or any solid malignancy that demonstrates an activating mutation in Harvey rat sarcoma viral oncogene homolog (HRAS), Kirsten rat sarcoma viral oncogene homolog (KRAS), or neuroblastoma RAS viral (v-ras) oncogene homolog (NRAS); Part 1 dose expansion (PD cohort[s]) and part 2: Advanced (metastatic or non-resectable) SCLC with any mutational status, or adenocarcinoma of the colon or rectum, or NSCLC or adenocarcinoma of the pancreas, all of which must demonstrate an activating mutation in HRAS, KRAS, or NRAS; Part 2 "basket" cohort: Advanced (metastatic or non-resectable) solid malignancy that demonstrates Ras pathway activation (including but not limited to activating BRAF/HRAS/KRAS/NRAS mutation, inactivating neurofibromin (NF1) mutation, or evidence of Ras pathway activation by gene expression analysis).
* Disease that did not respond to, or progressed after, at least 1 prior line of therapy, or has no generally-accepted standard therapy (dose escalation cohorts and optional "basket" cohort only).
* Measurable disease during part 1, measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1 is recommended but not required. Subjects enrolled in part 2 must demonstrate measurable disease per RECIST v1.1.
* PD expansion subjects only: Subjects must consent to pre-dosing and on-therapy tumor biopsies and additional sample collection procedures.
* All prior treatment-related toxicities must be National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v4 <=Grade 1 (except alopecia [permitted at any grade]) and peripheral neuropathy (permitted at <=Grade 2) at the time of screening.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1.
* Must have adequate organ function as defined by the following values: Absolute neutrophil count (ANC) >=1.5 x 10^9/liter (L); hemoglobin >=9 grams per deciliter (g/dL) subjects that required transfusion or growth factor need to demonstrate stable hemoglobin for 7 days of 9 g/dL; platelets >=100 x 10^9/L; prothrombin time (PT)/International normalized ration (INR) and partial thromboplastin time (PTT) <=1.5 x upper limit of normal (ULN); albumin >=2.5 g/dL; total bilirubin <=1.5 x ULN; aspartate transaminase (AST) <=2.5 x ULN; alanine transaminase (ALT) <=2.5 x ULN OR <5 x ULN; estimated glomerular filtration rate >=50 milliliter (mL)/minute/1.73 m^2; ejection fraction>= lower limit of normal (LLN); troponin <=ULN
* Able to swallow and retain orally administered medication.
* A female subject is eligible to participate if she is of: Non-childbearing potential; Childbearing potential and agrees to use one of the contraception methods from the time of the screening pregnancy test until at least 7 months after the last dose of study treatment; All female subjects of childbearing potential must have a negative serum pregnancy test <=7 days prior to first dose of study treatment; Female subjects who are lactating must discontinue nursing prior to the first dose of study treatment and must refrain from nursing throughout the treatment period and for 5 half-lives of GSK525762/trametinib or at least 28 days (whichever is longer) following the last dose of study treatment.
* Male subjects with female partners of childbearing potential must agree to abide by the reproductive guidelines from the first dose of study treatment and for at least 16 weeks after the last dose of study treatment.

Exclusion Criteria:

* Primary malignancy of the central nervous system or malignancies related to human immunodeficiency virus (HIV) or solid organ transplant.
* Prior therapy with any BET inhibitor.
* Recent prior therapy, defined as follows: Any non-biologic anti-cancer drug (either investigational or approved) within 14 days or 5 half-lives, whichever is longer, prior to the first dose of GSK525762 and trametinib; any nitrosoureas or mitomycin C within 42 days prior to the first dose of GSK525762 and trametinib; any biologic anti-cancer agent within 28 days prior to the first dose of GSK525762 and trametinib; any radiotherapy within 14 days or major surgery within 28 days prior to the first dose of GSK525762 and trametinib.
* Therapeutic-dose anticoagulation (e.g., warfarin, heparin) must be discontinued and coagulation parameters must be normalized prior to the first dose of GSK525762 and trametinib. Low dose (prophylactic) low molecular weight heparin or other anticoagulants are permitted.
* Current or planned use of a prohibited medication during treatment with GSK525762 and trametinib.
* Evidence of severe or uncontrolled systemic diseases (e.g., unstable or uncompensated respiratory, hepatic, renal, cardiac disease, or clinically significant bleeding episodes). Any serious and/or unstable pre-existing medical (aside from malignancy) condition, psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures, in the opinion of the investigator.
* Symptomatic or untreated leptomeningeal or brain metastases or spinal cord compression. Subjects with a history of central nervous system (CNS) involvement may be enrolled so long as all of the following requirements are met: Subjects must have received definitive therapy for the CNS involvement (e.g., surgery, radiotherapy, or stereotactic radiosurgery [i.e., gamma knife or equivalent]); At least 28 days must have elapsed since the CNS-directed therapy; All symptoms and AEs from the CNS-directed therapy must have resolved to <=Grade 1; Lesion stability must be demonstrated by serial imaging spaced at least 28 days apart; If the subject remains on corticosteroids, the dose must be stable to decreasing for the 28-day interval prior to study Day 1; The subject does not receive any enzyme-inducing anticonvulsants (EIACs) from 14 days prior to study Day 1 until the End of Treatment.
* Cardiac abnormalities as evidenced by any of the following: Baseline QTcF interval >450 millisecond (msec); Clinically significant conduction abnormalities or arrhythmias; Presence of cardiac pacemaker or defibrillator with a paced ventricular rhythm limiting ECG analysis; History or evidence of current >=Class II congestive heart failure as defined by New York Heart Association (NYHA); History of acute coronary syndromes (including unstable angina and myocardial infarction), coronary angioplasty, or stenting within the past 3 months. Subjects with a history of stent placement requiring ongoing antithrombotic therapy (e.g., clopidogrel, prasugrel) will not be permitted to enroll.
* Current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones, liver metastases, or otherwise stable chronic liver disease per investigator assessment).
* Presence of hepatitis B surface antigen (HBsAg) or positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment.
* History of known HIV infection or positive HIV test at screening.
* Any serious known immediate or delayed hypersensitivity reaction(s) to GSK525762 or trametinib, or idiosyncrasy to drugs chemically related to the investigational drugs.
* Subjects with a history of known bleeding disorder(s) or history of clinically significant (as judged by the investigator and medical monitor) hemorrhage (e.g., GI, neurologic, pulmonary) within the past 6 months.
* History of retinal vein occlusion.
* History of pneumonitis or interstitial lung disease.
* Any clinically significant gastrointestinal abnormalities that may alter absorption of oral medications, (e.g., malabsorption syndrome).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-11-27 (Estimated); Primary Completion 2020-08-19 (Estimated); Study Completion 2020-08-19 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of subjects with adverse events (AEs) and serious adverse events (SAEs) | Up to 12 months
  An AE is any untoward medical occurrence in a subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgement will be categorized as SAE.
Part 1: Number of subjects with dose limiting toxicities (DLT) as a measure of safety | Up to 12 months
  DLT is defined by the occurrence of severe toxicities during the first cycle of cancer therapy. An event will be considered a DLT if it occurs within the first 21 days of treatment and meets the DLT criteria.
Part 1: Area under the plasma concentration time curve from time 0 to last time of quantifiable concentration (AUC [0-T]) of GSK525762 and trametinib | Pre-dose,30minutes ±5minutes,1 hour±5minutes,2hours±10 minutes,3hours±10minutes, 4hours±15minutes,6±1hour,8±1hour, and 24±2hours at Day1 Week1;Day1 Week3. Pre-dose;1hour±10minutes post-dose at Day1 Week2,Day1 Week 4;every 8 Weeks from Week8 to Week52
  Blood samples will be collected at the indicated time points for pharmacokinetic analysis and concentration of GSK525762 and trametinib will be determined in plasma.
Part 1: Pre-dose (trough) concentration at the end of a dosing interval (Ctau) of GSK525762 and trametinib | Pre-dose,30minutes ±5minutes,1 hour±5minutes,2hours±10 minutes,3hours±10minutes, 4hours±15minutes,6±1hour,8±1hour, and 24±2hours at Day1 Week1;Day1 Week3. Pre-dose;1hour±10minutes post-dose at Day1 Week2,Day1 Week 4;every 8 Weeks from Week8 to Week52
  Blood samples will be collected at the indicated time points for pharmacokinetic analysis and concentration of GSK525762 and trametinib will be determined in plasma.
Part 1: Maximum observed plasma concentration (Cmax) of GSK525762 and trametinib | Pre-dose,30minutes ±5minutes,1 hour±5minutes,2hours±10 minutes,3hours±10minutes, 4hours±15minutes,6±1hour,8±1hour, and 24±2hours at Day1 Week1;Day1 Week3. Pre-dose;1hour±10minutes post-dose at Day1 Week2,Day1 Week 4;every 8 Weeks from Week8 to Week52
  Blood samples will be collected at the indicated time points for pharmacokinetic analysis and concentration of GSK525762 and trametinib will be determined in plasma.
Part 1: Time to Cmax (Tmax) of GSK525762 and trametinib | Pre-dose,30minutes ±5minutes,1 hour±5minutes,2hours±10 minutes,3hours±10minutes, 4hours±15minutes,6±1hour,8±1hour, and 24±2hours at Day1 Week1;Day1 Week3. Pre-dose;1hour±10minutes post-dose at Day1 Week2,Day1 Week 4;every 8 Weeks from Week8 to Week52
  Blood samples will be collected at the indicated time points for pharmacokinetic analysis and concentration of GSK525762 and trametinib will be determined in plasma.
Part 1: Change from Baseline in the phosphorylation of extracellular signal-regulated kinase (pERK) levels | Baseline and up to Week 3
  The pERK levels will be assessed in pre-therapy and on-therapy tumor samples.
Part 1: Change from Baseline circulating protein or ribonucleic acid (RNA) biomarkers | Baseline and up to Week 3
  The circulating protein or RNA biomarkers including to monocyte chemoattractant protein-1 (MCP-1) will be assessed in pre-therapy and on-therapy blood samples.
Part 1: Change from Baseline transcriptional levels and mitogen activated protein (MAP) kinase signaling | Baseline and up to Week 3
  The transcriptional levels and MAP kinase signaling will be assessed in pre-therapy and on-therapy tumor and/or blood samples.
Part 1: Overall response rate (ORR) | Up to 12 months
  ORR is defined as the percentage of subjects with a confirmed complete response (CR) or partial response (PR) at any time as per disease-specific criteria.
Part 1: Disease control rate (DCR) | Up to 12 months
  DCR is defined as the percentage of subjects with a confirmed CR, PR, or SD at any time as per disease-specific criteria.
Part 1: Duration of response (DOR) | Up to 12 months
  The DOR is defined as, in the subset of subjects who show a confirmed CR or PR, the time from first documented evidence of CR or PR until the first documented sign of disease progression or death.
Part 2: ORR | Up to 24 months
  ORR is defined as the percentage of subjects with a confirmed CR or PR at any time as per disease-specific criteria.
Part 2: Clinical response | Up to 24 months
  Clinical response is defined as confirmed ORR as per standard evaluation criteria. ORR is the percentage of subjects with a confirmed CR or PR at any time as per disease-specific criteria.
Part 2: Number of subjects with AEs and SAEs | Up to 24 months
  An AE is any untoward medical occurrence in a subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgement will be categorized as SAE.
Part 2: Number of subjects with dose reductions or delays as a measure of safety | Up to 24 months
  Dose reductions or delays will be evaluated until the end of treatment.
Part 2: Number of subjects withdrawals due to toxicities | Up to 24 months
  Withdrawals will be collected until the end of treatment.
Part 2: Number of subjects with abnormal clinical chemistry laboratory tests | Up to 24 months
  Clinical chemistry parameters will be analyzed as a measure of safety.
Part 2: Number of subjects with abnormal hematology laboratory tests | Up to 24 months
  Hematology parameters will be analyzed as a measure of safety.
Part 2: Number of subjects with abnormal routine urinalysis laboratory tests | Up to 24 months
  Urinalysis will be carried out as a measure of safety.
Part 2: Number of subjects with abnormal systolic blood pressure (SBP) and diastolic blood pressure (DBP) as a measure of safety | Up to 24 months
  Systolic and diastolic blood pressure will be measured in semi-supine position after 5 minutes of rest.
Part 2: Number of subjects with abnormal pulse rate | Up to 24 months
  Pulse rate will be measured in a semi-supine position after 5 minutes of rest..
Part 2: Number of subjects with abnormal respiratory rate | Up to 24 months
  Respiratory rate will be measured in a semi-supine position after 5 minutes of rest.
Part 2: Number of subjects with abnormal body temperature | Up to 24 months
  Body temperature will be measured in a semi-supine position after 5 minutes of rest.
Part 2: Number of subjects with abnormal electrocardiogram (ECG) findings | Up to 24 months
  Triplicate 12-lead ECGs will be obtained at each time point using an ECG machine to measure PR, QRS, QT, and Corrected QT interval (QTc).
Part 2: Number of subjects with cardiotoxicity and gastrointestinal (GI) toxicity | Up to 24 months
  Echocardiography (ECHO) or multigated acquisition (MUGA) scan will be performed to assess cardiotoxicity and GI effects will be monitored.
Part 2: AUC [0-T] of GSK525762 and trametinib | Pre-dose, and 0.5hour±5 minutes, 1-2 hours, 4-6hours post-dose at Day1 Week 1, Day1 Week3, and every 8 Weeks from Week8 to Week52
  Blood samples will be collected at the indicated time points for pharmacokinetic analysis and concentration of GSK525762 AND TRAMETINIB will be determined in plasma.
Part 2: Ctau of GSK525762 and trametinib | Pre-dose, and 0.5hour±5 minutes, 1-2 hours, 4-6hours post-dose at Day1 Week 1, Day1 Week3, and every 8 Weeks from Week8 to Week52
  Blood samples will be collected at the indicated time points for pharmacokinetic analysis and concentration of GSK525762 and trametinib will be determined in plasma.
Part 2: Cmax of GSK525762 and trametinib | Pre-dose, and 0.5hour±5 minutes, 1-2 hours, 4-6hours post-dose at Day1 Week 1, Day1 Week3, and every 8 Weeks from Week8 to Week52
  Blood samples will be collected at the indicated time points for pharmacokinetic analysis and concentration of GSK525762 and trametinib will be determined in plasma.
Part 2: Tmax of GSK525762 and trametinib | Pre-dose, and 0.5hour±5 minutes, 1-2 hours, 4-6hours post-dose at Day1 Week 1, Day1 Week3, and every 8 Weeks from Week8 to Week52
  Blood samples will be collected at the indicated time points for pharmacokinetic analysis and concentration of GSK525762 and trametinib will be determined in plasma.
Part 2: Change from Baseline in the pERK levels | Baseline and up to Week 3
  The pERK levels will be assessed in pre-therapy and on-therapy tumor samples.
Part 2: Change from Baseline circulating protein or RNA biomarkers | Baseline and up to Week 3
  The circulating protein or RNA biomarkers including to MCP-1 will be assessed in pre-therapy and on-therapy blood samples.
Part 2: Change from Baseline transcriptional levels and MAP kinase signaling | Baseline and up to Week 3
  The transcriptional levels and MAP kinase signaling will be assessed in pre-therapy and on-therapy tumor and/or blood samples.

SECONDARY OUTCOMES:
Part 1: Number of subjects with AEs and SAEs | Up to 12 months
  An AE is any untoward medical occurrence in a subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgement will be categorized as SAE.
Part 1: Number of subjects with dose reductions or delays as a measure of safety | Up to 12 months
  Subjects will be evaluated for dose reductions and delays. An event will be considered a DLT if it occurs within the first 21 days of treatment and meets the DLT criteria.
Part 1: Number of subject withdrawals due to toxicities | Up to 12 months
  DLT is defined by the occurrence of severe toxicities during the first cycle of cancer therapy. An event will be considered a DLT if it occurs within the first 21 days of treatment and meets the DLT criteria.
Part 1: Number of subjects with abnormal clinical chemistry laboratory tests | Up to 12 months
  Clinical chemistry parameters will be analyzed as a measure of safety.
Part 1: Number of subjects with abnormal hematology laboratory tests | Up to 12 months
  Hematology parameters will be analyzed as a measure of safety.
Part 1: Number of subjects with abnormal routine urinalysis laboratory tests | Up to 12 months
  Urinalysis will be carried out as a measure of safety.
Part 1: Number of subjects with abnormal SBP and DBP as a measure of safety | Up to 12 months
  Systolic and diastolic blood pressure will be measured in semi-supine position after 5 minutes of rest.
Part 1: Number of subjects with abnormal pulse rate | Up to 12 months
  Pulse rate will be measured in a semi-supine position after 5 minutes of rest.
Part 1: Number of subjects with abnormal respiratory rate | Up to 12 months
  Respiratory rate will be measured in a semi-supine position after 5 minutes of rest.
Part 1: Number of subjects with abnormal body temperature | Up to 12 months
  Body temperature will be measured in a semi-supine position after 5 minutes of rest.
Part 1: Number of subjects with abnormal ECG findings | Up to 12 months
  Triplicate 12-lead ECGs will be obtained at each time point using an ECG machine to measure PR, QRS, QT, and QTc.
Part 1: Number of subjects with cardiotoxicity and GI toxicity | Up to 12 months
  Echocardiography (ECHO) or multigated acquisition (MUGA) scan will be performed to assess cardiotoxicity and GI effects will be monitored.
Part 1: (AUC [0-T]) of GSK525762 and trametinib | Pre-dose,30minutes ±5minutes,1 hour±5minutes,2hours±10 minutes,3hours±10minutes, 4hours±15minutes,6±1hour,8±1hour, and 24±2hours at Day1 Week1;Day1 Week3. Pre-dose;1hour±10minutes post-dose at Day1 Week2,Day1 Week 4;every 8 Weeks from Week8 to Week52
  Blood samples will be collected at the indicated time points for pharmacokinetic analysis and concentration of GSK525762 and trametinib will be determined in plasma.
Part 1: Ctau of GSK525762 and trametinib | Pre-dose,30minutes ±5minutes,1 hour±5minutes,2hours±10 minutes,3hours±10minutes, 4hours±15minutes,6±1hour,8±1hour, and 24±2hours at Day1 Week1;Day1 Week3. Pre-dose;1hour±10minutes post-dose at Day1 Week2,Day1 Week 4;every 8 Weeks from Week8 to Week52
  Blood samples will be collected at the indicated time points for pharmacokinetic analysis and concentration of GSK525762 and trametinib will be determined in plasma.
Part 1: Cmax of GSK525762 and trametinib | Pre-dose,30minutes ±5minutes,1 hour±5minutes,2hours±10 minutes,3hours±10minutes, 4hours±15minutes,6±1hour,8±1hour, and 24±2hours at Day1 Week1;Day1 Week3. Pre-dose;1hour±10minutes post-dose at Day1 Week2,Day1 Week 4;every 8 Weeks from Week8 to Week52
  Blood samples will be collected at the indicated time points for pharmacokinetic analysis and concentration of GSK525762 and trametinib will be determined in plasma.
Part 1: Tmax of GSK525762 and trametinib | Pre-dose,30minutes ±5minutes,1 hour±5minutes,2hours±10 minutes,3hours±10minutes, 4hours±15minutes,6±1hour,8±1hour, and 24±2hours at Day1 Week1;Day1 Week3. Pre-dose;1hour±10minutes post-dose at Day1 Week2,Day1 Week 4;every 8 Weeks from Week8 to Week52
  Blood samples will be collected at the indicated time points for pharmacokinetic analysis and concentration of GSK525762 and trametinib will be determined in plasma.
Part 1: ORR | Up to 12 months
  ORR is defined as the percentage of subjects with a CR or PR at any time as per disease-specific criteria.
Part 1: DCR | Up to 12 months
  DCR is defined as the percentage of subjects with a confirmed CR, PR, or SD at any time as per disease-specific criteria.
Part 1: DOR | Up to 12 months
  The DOR is defined as, in the subset of subjects who show a confirmed CR or PR, the time from first documented evidence of CR or PR until the first documented sign of disease progression or death.
Part 1: Progression-free survival (PFS) | Up to 12 months
  PFS defined as the time from first dose of study treatment until the disease progression or death due to any cause.
Part 2: PFS | Up to 24 months
  PFS defined as the time from first dose of study treatment until the disease progression or death due to any cause.
Part 2: DOR | Up to 24 months
  The DOR is defined as, in the subset of subjects who show a confirmed CR or PR, the time from first documented evidence of CR or PR until the first documented sign of disease progression or death.
Part 2: DCR | Up to 24 months
  DCR is defined as the percentage of subjects with a confirmed CR, PR, or SD at any time as per disease-specific criteria.
Part 2 :Concentrations of GSK525762 and its relevant metabolite(s) and trametinib following repeat dose oral administration. | Pre-dose, and 0.5hour±5 minutes, 1-2 hours, 4-6hours post-dose at Day1 Week 1, Day1 Week3, and every 8 Weeks from Week8 to Week52
  Plasma samples will be collected at the indicated time points to measure concentrations of GSK525762 and its relevant metabolite(s) and trametinib following repeat dose oral administration.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline